CLINICAL TRIAL: NCT00149318
Title: Evaluation of the Long Term Efficacy of Enzyme Replacement Therapy in Fabry Disease
Brief Title: Enzyme Replacement Therapy in Fabry Disease
Status: Terminated | Type: Observational
Why Stopped: Difficulties in the patient's enrolment
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: FABRY DISEASE
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood on EDTA. Serum. Urine samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Fabry disease
  Interventions: Other: Biochemical analyses.

INTERVENTIONS:
Other: Biochemical analyses. — Biochemical analyses.

SUMMARY:
Fabry disease is an X-linked rare metabolic disease, caused by a deficient activity of the hydrolase α-Galactosidase A, and characterized by a progressive and systematic deposition of glycosphingolipids in many organs.

The disease is most severe in affected males. In the classic form (where the enzyme activity is absent) the clinical findings are represented by pain and paresthesias in the extremities, vessel ectasia (called angiokeratoma) in skin and mucous membranes, and hypohidrosis (a reduced sweating) during childhood or adolescence. Corneal and lenticular opacities may be present. Proteinuria, renal impairment,cardiac and neurological lesions develop with time, together with hypertension. When end stage renal disease occurs, dialysis or renal transplantation may be necessary. In heterozygous females a residual enzymatic activity may be demonstrated and they usually have asymptomatic or later onset disease manifestations, although rarely they could develop a disease as severe as in males.

A cardiac and a renal variant, where the heart and kidney are the only organs involved by the disease have been described too.

The recombinant human α-galactosidase A is now available for patients. Infusions of the enzyme replacement treatment have been demonstrated to be safe and effective. This study wants to evaluate the long term efficacy of enzyme replacement therapy in patients with Fabry disease and renal involvement.

Clinical period evaluations together with a genetic counselling will be offered to each patient.

DETAILED DESCRIPTION:
INTRODUCTION Fabry disease is an X-linked error of glycosphingolipid catabolism caused by the deficient activity of the lysosomal hydrolase α-galactosidase A (α-gal A) in tissues and fluids of affected hemizygous males; most heterozygous females have an intermediate level of enzymatic activity. The enzymatic defect leads to a systemic deposition of glycosphingolipids, predominantly globotriaosylceramide (Gb3), in body fluids and in the lysosomes of endothelial, perithelial, and smooth-muscle cells of blood vessels. Deposition also occurs in ganglion cells.

Clinical manifestations in classically affected hemizygotes (with absent α-gal A activity), include pain and paresthesias in the extremities, vessel ectasia (angiokeratoma) in skin and mucous membranes, and hypohidrosis during childhood or adolescence. Corneal and lenticular opacities are early findings. With increasing age, proteinuria and renal impairment lead to hypertension and uremia. Renal failure typically occurs in the third-fifth decades of life, and these patients need chronic hemodialysis and/or renal transplantation.

Atypical hemizygotes with residual α-gal A activity may be asymptomatic or have late-onset, mild disease manifestations primarily limited to the heart (the "cardiac variant"). Recently a renal variant has been identified too. Heterozygous females may have an attenuated form of the disease.The most frequent clinical finding in females is the characteristic whorl-like corneal epithelial dystrophy. They usually are asymptomatic, although rarely can be severely affected as hemizygous males.

In the kidney accumulation of glycosphingolipids appear in the sequence in endothelial and epithelial cells of the glomerulus and of Bowman's space, epithelium of the loops of Henle and in distal tubules till proximal tubules, interstitial histiocytes and fibrocytes. Lipid-laden distal tubular epithelial cells desquamate and may be detected in the urinary sediment.

Renal blood vessels may be involved progressively and extensively. An early finding is arterial fibrinoid deposits. Other histologic renal findings are severe arteriolar sclerosis, glomerular atrophy and fibrosis, pseudotubular proliferation of residual glomerular epithelium, tubular atrophy and diffuse interstitial fibrosis. Preliminary studies of enzyme replacement therapy demonstrate that periodic infusions of recombinant human α-galactosidase A are safe and effective in patients with Fabry disease.

The purpose of this study is to evaluate the long term efficacy of enzyme replacement therapy in patients with Fabry disease and renal involvement.

AIM Primary

* To evaluate the effect of enzyme replacement therapy on the rate of decline in the glomerular filtration rate (GFR, measured by inulin clearance) in Fabry patients with renal involvement
* To evaluate the biological activity of recombinant human galactosidase in terms of clearance of plasma Gb3 (that is directly correlated with renal endothelial glycosphingolipid clearance) Secondary

To evaluate the effect of enzyme replacement therapy on:

* 24-hour urinary protein excretion
* renal plasma flow (PAH renal clearance)
* glomerular perm-selectivity (fractional dextran clearances)
* end stage renal failure, kidney transplantation or death
* systolic and diastolic blood pressure
* cardiac anomalies (left ventricular hypertrophy, arrhythmias, conduction anomalies)
* cutaneous anomalies
* ocular anomalies DESIGN Twenty patients (males and females) with Fabry disease, and renal involvement, referred to the SMIMAF - Studio Multicentrico Italiano sulla Malattia di Anderson-Fabry - will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 16 years and ≤ 65 years
* clinical diagnosis of Fabry disease, confirmed by α-galactosidase A assay and detection of mutation in α-GalA gene
* serum creatinine ≥ 1.4 mg/dl (females) and ≥ 1.6 mg/dl (males) and/or proteinuria ≥ 0.4 g/24h
* written informed consent

Exclusion Criteria:

* any clinically relevant condition that may affect study participation and/or study results
* inability to fully understand the purpose and the risks of the study

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Fabry disease.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2002-12; Primary Completion 2008-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Daina, MD, Principal Investigator — Mario Negri Institute
Locations (1):
- Clinical Research Center for Rare Diseases, Ranica, Bergamo, Italy